CLINICAL TRIAL: NCT01031329
Title: Identification and Characterization of the Bacteria Causing Acute Otitis Media (AOM) Episodes in Young Children in Turkey
Brief Title: Study to Identify and Characterize Bacteria Causing Acute Otitis Media in Young Children in Turkey
Status: Withdrawn | Type: Observational
Why Stopped: Key aspects linked to sample management and analysis were not met during feasibility assessment limiting the ability of the study to reach its objectives.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111339
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Infections, Streptococcal
MeSH Terms: conditions — Streptococcal Infections | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Middle ear fluid and urine.

GROUPS / COHORTS (1):
- Complicated Acute otitis media Group: This group was divided into 3 sub-groups.
  * One sub-group includes treatment failure subjects who have had a diagnosis of acute otitis media and showed no clinical improvement within 48-72 hours of antibiotic treatment or reappearance of symptoms within 10 days following the end of antibiotic treatment.
  * The second sub-group includes subjects with recurrent acute otitis media, who have had new episodes of acute otitis media within the past 6 months or the fourth (or greater) new episode within the past year.
  * The third sub-group includes subjects with spontaneous otorrhoea if perforation has occurred < 24 hours prior to the visit.
  Interventions: Procedure: Tympanocenthesis and urine collection

INTERVENTIONS:
Procedure: Tympanocenthesis and urine collection — Fluid using needle aspiration is obtained from middle ear fluid. Urine is collected using a urine bag.

SUMMARY:
The purpose of this study is to identify and characterize the bacteria causing complicated Acute Otitis Media episode in children >= 3 months to < 5 years in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Age: >= 3 months and < 5 years at the time they are seen by the paediatrician. The subject becomes ineligible on the fifth birthday.
* Signs, symptoms, and conditions:
* One of the functional or general signs of otalgia ,conjunctivitis, fever and either
* Paradise's criteria or
* Spontaneous otorrhoea of less than 24 hours.
* Subjects if classified as recurrent acute otitis media or treatment failure as described below:
* Recurrent acute otitis media: Defined as a subject who has an episode of acute otitis media representing the third new episode within the past 6 months, or the fourth new episode within the past year.
* Treatment failure: Defined as a subject who was diagnosed with acute otitis media and received antibiotic treatment from a physician, but is still symptomatic 48-72 hours after initiation of the treatment. As with other acute otitis media cases, the onset of signs or symptoms should have been within 72 hours prior to the initial visit to the physician.
* Written informed consent obtained from parent or guardian prior to study start.

Exclusion Criteria:

* Hospitalised during the diagnosis of acute otitis media or during treatment.
* Otitis externa, or otitis media with effusion.
* Presence of a transtympanic aerator.
* Systemic antibiotic treatment received for a disease other than acute otitis media in the 72 hours prior to enrolment.
* Receiving antimicrobial prophylaxis for recurrent acute otitis media.
* Provision of antibiotic by paediatrician at the enrolment visit prior to the sampling of the middle ear fluid or spontaneous otorrhoea.
* Patients that are on antibiotics for acute otitis media, and are clinically improving.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects aged >= 3 months and < 5 years, diagnosed as having complicated acute otitis media on routine clinical care in the study hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of bacterial pathogens isolated from middle ear fluid samples.

SECONDARY OUTCOMES:
Occurrence of bacterial serotypes.
Antimicrobial susceptibility of bacteria isolated from middle ear fluid samples collected from sub-groups of complicated acute otitis media cases.
Occurrence of treatment failure of acute otitis media and of recurrent acute otitis media.
Occurrence of bacteria in acute otitis media cases vaccinated with a pneumococcal vaccine.
Occurrence of spontaneous otorrhoea.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Turkey (Türkiye) (4):
  - GSK Investigational Site, Adana
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir